CLINICAL TRIAL: NCT01706887
Title: Clinical, Pharmacological and Biological Investigations of a Polymorphism of Nedd4 , a Regulatory Protein of the Epithelial Sodium Channel
Brief Title: Genetic Determinant of Blood Pressure Sensitivity to Salt Intake
Acronym: JEU004
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end of recruitment period was reach
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P060215
Record Dates: First submitted 2012-04-27; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-03

CONDITIONS: Hypertension
Keywords: Nedd4-2; blood pressure; polymorphism; salt intake; between 18 and 35 years old; BMI between 18 and 28 Kg per m2; no active disease; no alcool or drug abuse or smoke
MeSH Terms: conditions — Hypertension; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diet Amiloride (Experimental): One week Low Na diet (10 mmol/d) followed by ine week high Na diet (200 mmol/d) followed by 2 weeks administration of amiloride (10 mg the 1 st week and the 20mg).
  Interventions: Other: Diet Amiloride

INTERVENTIONS:
Other: Diet Amiloride — only arm of the trial

SUMMARY:
Nedd4.2 is a regulator of ENac, a transporter of sodium involved in the regulation of salt retention by the kidney. The study address the consequence of a frequent genetic variation leading expected to impact the function of Nedd4 and in turn, the ability of kidneys to excrete salt intake. Our hypothesis is that the genetic variants of Nedd4.2 could constitute a genetic predisposition to (or protection against) salt-sensitive hypertension.

DETAILED DESCRIPTION:
Subjects were submitted one week to a low sodium-high potassium diet, and then switch to a high sodium,-low potassium diet for two weeks. the last week, subject were taken a 20 MG daily dose of amiloride, a potassium sparing diuretic.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* between 18 and 35 years odl
* BMI between 18 and 28 Kg per m2
* non smokers
* no active disease
* no alcool or drug abuse

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Difference in Blood Pressure among genotypes | 24h AMBP will be measured weekly for the duration of study, an expected average of 3 weeks
  24h AMBP will be measured weekly for the duration of study, an expected average of 3 weeks

SECONDARY OUTCOMES:
Ambulatory Blood Pressure (AMBP) | three weeks
  24h AMBP was measured fourth : at the beginning of the study,at the end of the low sodium-high potassium diet, after one week under the high sodium-low potassium diet and at the end of amiloride treatment under high sodium-low potassium diet

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jeunemaître, PD, PhD, Principal Investigator — genetic department